CLINICAL TRIAL: NCT02157467
Title: The Effect of Coadministration of BMS-955176 on the Pharmacokinetics of a Combined Oral Contraceptive Containing Ethinyl Estradiol and Norgestimate in Female Subjects
Brief Title: Study of Combined Oral Contraceptive Effects in Female Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: ViiV Healthcare (Industry)
Collaborators: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 206293; AI468-041 (Other: Bristol-Myers Squibb)
Record Dates: First submitted 2014-06-02; First posted 2014-06-06 (Estimated); Last update posted 2018-04-17 (Actual); Status verified 2018-04

CONDITIONS: Infection, Human Immunodeficiency Virus
MeSH Terms: conditions — Infections; Acquired Immunodeficiency Syndrome | interventions — BMS-955176; Moxifloxacin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Arm 1: NGMN/EE + BMS-955176 (Experimental): Cycle 1- Active Ortho Cyclen QD on Days 1 to 21. Inert Ortho Cyclen tablets on Days 22 to 28
  Cycle 2- Active Ortho Cyclen QD alone on Days 29 to 39 (11 days), followed by concomitant administration of active Ortho Cyclen QD + BMS-955176 80 mg QD on Days 40 to 49 (10 days)
  Interventions: Drug: BMS-955176; Drug: Ortho Cyclen

INTERVENTIONS:
Drug: BMS-955176
Drug: Ortho Cyclen

SUMMARY:
The purpose of this study is to assess the effect of BMS-955176 on the pharmacokinetics of coadministered oral contraceptives.

ELIGIBILITY:
Inclusion Criteria:

1. Signed Written Informed Consent a) The signed informed consent form
2. Target population

   * a) Healthy female subjects as determined by no clinically significant deviation from normal in medical history, physical examination findings, vital sign measurements, 12-lead ECG measurements, physical measurements, and clinical laboratory test results
   * b) Body Mass Index (BMI) of 18.0 to 32.0 kg/m2, inclusive, at screening and Day -1. BMI = weight (kg)/[height (m)]2
   * c) Weight greater than or equal to 45 kg
   * d) Subject Reenrollment: This study permits the reenrollment of a subject that has discontinued study as a pretreatment failure (ie, has not been treated). If reenrolled, the subject must be reconsented
3. Age and Reproductive Status

   * a) Women, 18 to 40 years of age, inclusive
   * b) Women of childbearing potential (WOCBP) with intact ovarian function as determined by medical history and history of regular menstrual cycles, and who have been on a stable regimen of Ortho Cyclen for at least 2 consecutive months without evidence of breakthrough bleeding or spotting, or subjects who have been using a stable regimen of another combination oral contraceptive containing EE for at least two months prior to dosing on Day 1 of Cycle 1 and willing to switch to Ortho Cyclen for the total duration of the study (approximately 78 days)
   * c) Women must have a negative serum or urine pregnancy test (minimum sensitivity 25 IU/L or equivalent units of human chorionic gonadotropin) within 24 hours prior to dosing on Day 1 of Cycle 1
   * d) Women must not be breastfeeding

Exclusion Criteria:

Medical History and Concurrent Diseases

* a) Any significant acute or chronic medical illness
* b) History of biliary disorders, including Gilbert's disease or Dubin-Johnson disease
* c) Current or recent (within 3 months of dosing on Day 1 of Cycle 1) gastrointestinal disease
* d) Any major surgery within 4 weeks of dosing on Day 1 of Cycle 1
* e) Any gastrointestinal surgery (including cholecystectomy) that could impact upon the absorption of study drug
* f) Donation of > 400 mL to a blood bank or in a clinical study (except a screening visit) within 8 weeks of dosing on Day 1 of Cycle 1
* g) Blood transfusion within 4 weeks of dosing on Day 1 of Cycle 1
* h) Inability to tolerate oral medication
* i) Inability to be venipunctured and/or tolerate venous access
* j) Smokers (those who currently smoke, as well as those who have stopped smoking less than 6 months prior to dosing on Day 1 of Cycle 1)
* k) Recent (within 6 months of dosing on Day 1 of Cycle 1) drug or alcohol abuse as defined in Diagnostic and Statistical Manual of Mental Disorders, fourth edition (DSM IV), Diagnostic Criteria for Drug and Alcohol Abuse
* l) Any other sound medical, psychiatric, and/or social reason as determined by the investigator

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 46 (Actual)
Dates: Start 2014-06-02 (Actual); Primary Completion 2014-08-25 (Actual); Study Completion 2014-08-25 (Actual)

PRIMARY OUTCOMES:
Serial blood samples for plasma Ethinyl Estradiol and Norelgestromin determination | Before dosing (0 hour) through 24 hours after administration on Days 21 and 49

SECONDARY OUTCOMES:
Serum progesterone measurements | Day 14, 21, 35, and 42
Trough blood samples collected for BMS-955716 | Days 48, 49, 50
Safety assessments based on review of adverse events, vital sign measurements, electrocardiograms, physical examinations, and clinical laboratory tests. | Two to three months

CONTACTS AND LOCATIONS:
Overall Officials: Viiv Clinical Trials, Study Director — ViiV Healthcare